CLINICAL TRIAL: NCT06144450
Title: Evaluation of Effectiveness of the Web-Based Monitoring Program Given to Mothers of Premature Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rukiye Çelik, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-439
Record Dates: First submitted 2023-11-01; First posted 2023-11-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Infant Development; Maternal Stress; Growth
Keywords: premature infant; mother; discharge; transition to home; home care; nurse
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The presented modules will be made accessible to mothers in the experimental group through a website. The modules will be completed in order and the necessary forms and follow-ups will be completed at the end of each module.
  Interventions: Other: Web-Based Monitoring Program
- Control Group (No Intervention): No intervention will be made in the control group.

INTERVENTIONS:
Other: Web-Based Monitoring Program — The research will be carried out in three stages; (1) creating the content of the follow-up program, (2) designing the web page, (3) implementing the program with mothers. The topics to be included in the monitoring program will be prepared within the framework of the "Empowerment Model". Knowledge and attitude-self-efficacy will be tried to be increased with the modules to be prepared. Accordingly, the program is planned to consist of 3 modules. These are "Preparation for Hospital Discharge Module", "Transitional Care Module" and "Home Care Module". The presented modules will be made accessible to mothers in the experimental group through a website. The modules will be completed in order and the necessary forms and follow-ups will be completed at the end of each module.
  Arms: Intervention Group

SUMMARY:
The study was planned to determine the effect of the web-based hospital and home follow-up program given to mothers of premature infants on infant growth-development, repeated hospitalization of the infant, maternal stress, preparation for discharge, home care and problem-solving care skills. The population of the study will consist of mothers of premature infants receiving care and treatment in the neonatal intensive care units where the study is planned to be conducted between December 15, 2023 and December 01, 2024. Because no similar study was found in the literature, the sample calculation was performed using the G*power 3.1.9.2 program with effect size = 0.40, type 1 error = 0.05, and 95% power. The analysis yielded a sample size of 52, and considering a 20% loss rate, the total sample size was determined to be 62. Premature infants and their mothers sampled in the study will be assigned to the intervention and control groups by randomization with the stratified block method according to the gestation week, gender and birth weight of the infants. Block randomization will be done by creating 6 blocks consisting of 4 letters. Block randomization will be done by an academic independent of the research. The group with which the study will start will be determined by lottery by the independent academic and the participants will be assigned to the intervention and control groups with randomization envelopes. Mother Descriptive Information Form, Infant Descriptive Information and Follow-up Form, Preparation for Discharge from the Neonatal Intensive Care Unit and Home Care Scale, Neonatal Intensive Care Unit Parental Stress Scale, Problem Solving Skills Assessment Form, Ankara Developmental Screening Inventory, and Process Evaluation Form will be used for data collection. The research will be carried out in three stages; (1) creating the content of the follow-up program, (2) designing the web page, (3) implementing the program with mothers. The implementation of the program based on the Empowerment Model will be implemented in 3 stages: preparation of the premature infant hospitalized in the neonatal intensive care unit for discharge from the hospital, transition to home and home care.

DETAILED DESCRIPTION:
Premature infants' hospital, home transition, and home care needs differ from those of other infants. After being discharged from the neonatal intensive care unit, mothers become the primary caregivers for their premature infants at home. Therefore, discharge preparation should begin when the infant is admitted to the hospital, continue throughout the neonatal intensive care unit stay, and be supported by home follow-up. It has been observed that mothers who have not adequately prepared for discharge often find themselves unprepared for their infants' discharge from the hospital and for providing adequate care at home Nurses provide discharge preparation to facilitate the mother's preparation for discharge, the mother and infant's transition to home, and home care. This preparation can support the mother's stress level and problem-solving skills, as well as the infant's physiological stability and age-appropriate growth and development. Supporting and empowering mothers of premature infants while their infants are in the neonatal intensive care unit is a critical nursing intervention. Therefore, neonatal intensive care unit nurses can use the Family-Centered Empowerment Model to empower mothers. The Family-Centered Empowerment Model has been shown to increase parenting responsibility, care skills, parental self-efficacy, self-, quality of life, and emotional regulation, and to decrease the burden of care in mothers of sick children through integrated programs. The use of technology in healthcare makes information more accessible.

ELIGIBILITY:
Inclusion Criteria:

* For mothers

  * Those over 18 years of age,
  * Literate,
  * Having a computer or mobile phone,
  * Having access to internet connection,
  * Able to use the Internet,
  * Able to speak Turkish,
  * Primiparous,
  * Mothers who agree to participate in the study will be included in the study.
* For babies

  * 28-316. born during the week of pregnancy,
  * Birth weight 1000-2000 grams. the one which,
  * Hospitalized for at least 5 days,
  * Prematurity and related health problems (respiratory distress syndrome, intra cranial hemorrhage, patent ductus arteriosus, intrauterine growth retardation, small for gestational age, SEPSIS, retinopathy of prematurity, cholestasis, nutritional intolerance)
  * Babies without congenital anomalies will be included in the study.

Exclusion Criteria:

* Mothers with physical and/or mental disabilities,
* Mothers diagnosed with a psychological disease (severe depression, suicide attempt, etc.),
* Mothers who are addicted to alcohol and substances,
* Mothers who cannot complete the modules will not be included in the research.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Baby Monitoring Form -1 | at birth, 1st month, 3rd month
  Growth-development parameters of birth, discharge and home care (Height - meters)
Neonatal Intensive Care Unit Parental Stress Scale | at birth; through birth, an average of 3 months; through discharge, an average of 3 day; through discharge, an average of 3 month. (Increase and decrease over time will be evaluated.)
  Scale; The sub-dimensions are Babies' Appearance and Behavior, Sights and Sounds, Your Relationship with Your Baby, and Your Role as a Parent.
Problem Solving Skills Evaluation Form | at birth; through birth, an average of 3 months; through discharge, an average of 3 day; through discharge, an average of 3 month
  Subscales of the form are Child (Baby) Care Skill Subscale, Scanning Subscale, Formulation Subscale, Pre-evaluation (Prediction) Subscale, Planning Subscale, Application Subscale, Evaluation Subscale, Problem Solving Process Subscale.The lowest score that can be obtained from the entire scale is 27 and the highest score is 261.As the score increases, mothers' problem-solving skills increase.
Preparation for Discharge from Neonatal Intensive Care Unit and Home Care Scale | at birth; through birth, an average of 3 months; through discharge, an average of 3 day; through discharge, an average of 3 month
  The scale developed for mothers includes 4 sub-dimensions (feeding, general condition perception, hygienic care, care practices). A minimum of 22 and a maximum of 154 points can be obtained from the mother scale. High scores indicate that parents are ready for discharge.
Process Evaluation Form | through discharge, an average of 3 month
  9 open-ended questions are asked about the benefits of the program, satisfaction levels with the program, the effects of the program on the feeling of knowledge and competence in baby care, the conveniences and difficulties of the program, and suggestions for the program.This form is a form in which qualitative and quantitative data are collected. Therefore, it has no upper and lower scores.
Ankara Developmental Screening Inventory | through discharge, an average of 1 month; through discharge, an average of 3 month
  It is a screening inventory that provides in-depth and systematic information about the development of babies and children (0 -6 years old).The inventory consists of 4 subdomains: language-cognitive, fine motor, gross motor and social skills-self-care.
Baby Monitoring Form -2 | at birth, 1st month, 3rd month
  receiving emergency healthcare services after discharge (rate)

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye Çelik, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)